CLINICAL TRIAL: NCT02118415
Title: Targeted Natural Killer (NK) Cell Based Adoptive Immunotherapy for the Treatment of Patients With Non-Small Cell Lung Cancer (NSCLC) After Radiochemotherapy (RCT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSCLC-TKD/IL-2; 2008-002130-30 (EudraCT Number)
Record Dates: First submitted 2014-02-25; First posted 2014-04-21 (Estimated); Last update posted 2024-04-17 (Actual); Status verified 2023-11

CONDITIONS: NSCLC Stage IIIA/B
Keywords: not eligible for surgery; efficacy of immunotherapy following RCTx
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Participants of the intervention group receive biological product (ex vivo activated, autologous NK cells), participants of the control group receive no biological product
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventional (Experimental): Interventional group: activated autologous NK cells as a drug
  Interventions: Other: Hsp70-peptide TKD/IL-2 activated, autologous NK cells
- Control group (No Intervention): Control group: BSC

INTERVENTIONS:
Other: Hsp70-peptide TKD/IL-2 activated, autologous NK cells — Adjuvant treatment with Hsp70-peptide TKD/IL-2 activated, autologous NK cells following completion of standard radiochemotherapy (Cisplatin/Vinorelbine)
  Arms: Interventional

SUMMARY:
Targeted Natural Killer (NK) cell based adoptive immunotherapy for the treatment of patients with Non-Small Cell Lung Cancer (NSCLC) after radiochemotherapy (RCT)

DETAILED DESCRIPTION:
Patients with non-small cell lung carcinoma (NSCLC) in stage III A and III B showing at least stable disease after RCTx will be enrolled into the clinical trial. The aim of the study is to show the efficacy of an adjuvant treatment with Hsp70-peptide TKD/IL-2 activated, autologous NK cells following completion of standard radiochemotherapy (Cisplatin/Vinorelbine). Patients will be randomized 1:1 either to the interventional study group to receive 4 cycles of autologous immunotherapy with activated NK cells or to the control group (BSC).

ELIGIBILITY:
Inclusion Criteria:

* First diagnosis of histologically and/or cytologically proven and unresectable NSCLC with clinically stage III A and III B
* Completion of radiochemotherapy no longer than 8 weeks ago
* Progression free according to RECIST criteria at the first assessment after completion of RCTx
* Confirmed presence of Hsp70 on patient´s tumors
* ECOG Status(Appendices) ≤ 2

Exclusion Criteria:

* Any severe heart disease or any severe concomitant disease (ECOG stage > 2)
* NSCLC patients (stage IIIA/B) eligible for initial surgery with a confirmed consent of an interdisciplinary tumorboard
* Patients that show ALK positivity or an activating mutation of the EGFR-TK domain
* Patients with locally advanced or metastatic non-small cell lung cancer other than predominantly squamous cell histology
* Receipt of immunosuppressive drugs including high dose systemic corticosteroids within 3 weeks before study entry. Low dose corticosteroids as they are a common treatment option for patients suffering from COPD are not an exclusion criterium

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-03; Primary Completion 2018-03-28 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Progress free survival | follow up after randomization for at least 18 months

SECONDARY OUTCOMES:
overall survival (OS) | follow up after randomization for at least 18 months
toxicity (AE and SAE) | follow up after randomization for at least 18 months
quality of life (QoLQ-30, LC-13) | follow up after randomization for at least 18 months
biological parameters (NK cell activation) | follow up after randomization for at least 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum rechts der Isar, Strahlentherapie und Radiologische Onkologie, Munich, Germany